CLINICAL TRIAL: NCT07382440
Title: Observational Prospective Study to Evaluate Effectiveness of Subcutaneous Treatment With Foslevodopa/Foscarbidopa in Real Life Setting for Advanced Parkinson's Disease Patients in Belgium.
Brief Title: A Study to Assess Change in Disease Symptoms in Adult Participants With Advanced Parkinson Disease Using Subcutaneous Foslevodopa/Foscarbidopa in Belgium
Acronym: ProParkB
Status: Not yet recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P26-053
Record Dates: First submitted 2026-01-27; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease: Advanced Parkinson's Disease; Foslevodopa/Foscarbidopa
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Foslevodopa/Foscarbidopa: Participants will receive Foslevodopa/Foscarbidopa as prescribed by their physician according to local label.

SUMMARY:
Parkinson's disease (PD) is a neurological condition, which affects the brain. PD gets worse over time, but how quickly it progresses varies a lot from person to person. Some symptoms of PD are tremors, stiffness, and slowness of movement. This study will assess how effective Foslevodopa/Foscarbidopa is in treating adult participants with advanced Parkinson Disease under routine clinical practice in Belgium.

Foslevodopa/Foscarbidopa is an approved drug for the treatment of Parkinson's Disease. Approximately 120 adult participants who are prescribed Foslevodopa/Foscarbidopa by their doctors will be enrolled at 15 sites across Belgium.

Participants will receive Foslevodopa/Foscarbidopa subcutaneous infusion as prescribed by their physician. Participants will be followed for up to 18 months.

There is expected to be no additional burden for participants in this trial. Participants will attend regular visits during the study at a hospital or clinic according to their routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Participant diagnosed with Advanced Parkinson's Disease (PD), aged 18 years or older able to provide voluntary informed consent.
* Participant evaluated for commercially available continuous subcutaneous Foslevodopa/Foscarbidopa (LDp/CDp) in the hospital at the clinician's discretion as part of his/her routine clinical care and the intention to administer subcutaneous LDp/CDp made prior to and independent of recruitment into the study.

Exclusion Criteria:

* Participant participating in an interventional research study (not including noninterventional studies) during the administration of LDp/CDp.
* Participant evaluated for commercially available continuous subcutaneous LD/CDp outside of the hospital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with advanced Parkinson's Disease receiving Foslevodopa/Foscarbidopa treatment in accordance with the local label requirements in Belgium.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-01-28 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in OFF Time (hours) as measured by modified Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) IV | Up to approximately 6 months
  The Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is an investigator-used rating tool to follow the longitudinal course of Parkinson's Disease (PD)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=P26-053